CLINICAL TRIAL: NCT05840835
Title: A Phase 1/2a Open-Label, Dose-Escalation/Dose-Expansion Safety, Tolerability and Anti-tumor Activity Study of IMX-110 in Combination With Tislelizumab in Patients With Advanced Solid Tumors
Brief Title: Study of IMX-110 in Combination With Tislelizumab in Patients With Advanced Solid Tumors
Acronym: IMMINENT-01
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immix Biopharma, Inc. (Industry)
Collaborators: BeiGene (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMX-110-002
Record Dates: First submitted 2023-01-04; First posted 2023-05-03 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- IMX-110 in Combination With Tislelizumab (Experimental): Patients with advanced solid tumors will be administered a combination of IMX-110 with Tislelizumab
  Interventions: Drug: IMX-110 combined with Tislelizumab

INTERVENTIONS:
Drug: IMX-110 combined with Tislelizumab — Study of IMX-110 in Combination With Tislelizumab in Patients With Advanced Solid Tumors
  Other Names: One Arm

SUMMARY:
Phase 1/2a Phase 1 is an open-label, multicenter dose escalation/dose expansion study designed to assess the safety, tolerability, pharmacokinetics (PK) and antitumor activity of IMX-110 in combination with Tislelizumab. The recommended Phase 2 dose (RP2D) will be evaluated in further dose expansion Phase 2a study submitted as an amendment to this Phase 1 protocol during the conduct of the Phase 1 study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who are 16 years or older
* Patients with confirmed advanced solid tumor as per histology, who have progressed, are refractory, or are intolerant to standard therapy appropriate for tumor type
* Patients with an Eastern Cooperative Oncology Group (ECOG) Performance status of 0-2 (Appendix 2)
* Patients with a life expectancy of at least 3 months
* Patients with adequate cardiac function as measured by left ventricular ejection fraction >50%
* Patients who have not reached a cumulative total lifetime maximum dose of 550 mg/m2 doxorubicin or per investigator discretion
* Patients who meet the following laboratory requirements:
* Absolute neutrophil count (ANC) ≥ 1.0 x 109/L
* Hemoglobin (HGB) ≥ 9.0 g/dL (patients may be transfused to achieve this HGB level)
* Platelet count ≥ 100 x 109/L
* Total bilirubin level ≤ 1.5 x ULN, or ≤ 3.0 x ULN for patients with Gilbert syndrome
* AST and ALT ≤ 2.5 x ULN (≤5 x ULN if liver metastasis present)
* Creatinine ≤ 1.5 x ULN (Creatinine clearance >50 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal) (Creatinine clearance will be measured based on Cockcroft-Gault Equation).
* Women of childbearing potential and men must agree to sexual abstinence or to use highly effective, double barrier contraception during the study and for 6 weeks following the final dose of IMX-110. Double barrier contraception is defined as a condom AND one other form of the following:
* Birth control pills (The Pill)
* Depot or injectable birth control
* IUD (Intrauterine Device)
* Birth control patch (e.g. Ortho Evra)
* NuvaRing®
* Documented evidence of surgical sterilization at least 6 months prior to the screening visit, i.e., tubal ligation or hysterectomy for women or vasectomy for men.

Male patients must not donate sperm for at least 24 weeks post-dose of the last study treatment.

Females of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1.

Rhythm methods during the study and for 4 months after the dose of IMX-110 + Tislelizumab will not be acceptable.

Exclusion Criteria:

* Patients with a history of severe allergic reactions to any unknown allergens or any components of the study drug formulation.
* Patients receiving any chemotherapy within 14 days of dosing, immunotherapy within 28 days of dosing, or biologic or hormonal therapy within 28 days of dosing for cancer treatment (exclusively). Patients with prostate cancer can continue administration of Gonadotropin-releasing hormone (GnRH) agonists.
* Subject participating in any other drug study ≤ 4 weeks (6 weeks for immunotherapy investigational agents) or 5 half-lives of the investigational product, whichever is longer, prior to study drug administration or is scheduled to receive one during the treatment or post-treatment period.
* Patients who are expected to need surgery or benefit from other anti-cancer therapy to be initiated during the study period.
* Patients with a history of and/or risk factors for ischemic heart disease, congestive heart failure, symptomatic bradycardia, atrioventricular (AV) block of second degree or higher grade, prolonged QTcF interval (>450 msec in men and >470 msec in women and additional risk factors for QT prolongation (e.g. hyperthyroidism, electrolyte imbalance). (Pacemaker is not prohibited).
* Patients who have not recovered from adverse events (AEs; ≥ CTCAE grade 2) due to prior treatment (i.e. chemotherapy, targeted therapy, radiation, or surgery) within 7 days prior to Cycle 1 Day 1, unless deemed to be irreversible, or approved by the Sponsor and Medical Monitor.
* Females who are pregnant or lactating or intend to become pregnant before, during, or within 24 weeks after participating in this study; or intending to donate ova during such time period.
* Patients with a known positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C antibodies (HCV). Patients may be enrolled if they have HBV, HCVor HIV with viral load suppressed by anti-virals.

Any condition that, in the opinion of the investigator or sponsor, would interfere with evaluation of the investigational product.

* Active autoimmune diseases or history of autoimmune diseases that may relapse or history of life-threatening toxicity related to prior immune therapy. Note: Patients with the following diseases are not excluded and may proceed to further screening:
* Controlled type I diabetes (insulin dependent)
* Hypothyroidism (provided it is managed with hormone replacement therapy only)
* Controlled celiac disease
* Skin diseases not requiring systemic treatment (eg, vitiligo, psoriasis, alopecia)
* Any other disease that is not expected to recur in the absence of external triggering factors (requires consultation with the medical monitor prior to enrollment)
* Indicated live vaccines should be given ≥4 weeks prior to enrollment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-01-24 (Estimated); Study Completion 2024-01-24 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | 28 days
  Incidence, severity and causality of AE and serious adverse events (SAE) / Physical examination changes from baseline / Vital sign changes from baseline (heart rate, systolic/diastolic blood pressure, respiratory rate, and temperature) / Hematology and chemistry parameter changes from baseline / 12-lead ECG and 2-D Echocardiogram changes from baseline
Maximum tolerated doses (MTDs) and RP2D of IMX-110 in combination with Tislelizumab | 28 days
  MTD is defined as the highest dose at which ≤ 33% of the patients treated during the 3+3 design experience a DLT and/or at least two ≥ grade 2 non-hematologic toxicities during the first treatment cycle, and will be used to identify the RP2D to be taken forward to Phase 2a.

SECONDARY OUTCOMES:
Plasma concentrations of IMX-110 | 7 days
  Plasma concentration of IMX-110 will be measured when administered in treatment Cycle 1. Samples will be collected on Day 1 (pre-dose, and immediately after, 5 minutes, 1 hour, 1.5 hours, 3 hours, 5 hours post-dose), on Day 2 (pre-dose), and Day 5 (pre-dose and immediately after, 5 minutes, 1 hour, 1.5 hours, 3 hours, 5 hours post-dose), and optionally on Day 7 (pre-dose, 5 minutes, 15 minutes, 1 hour, 1.5 hours, 3 hours, 5 hours post-dose).
Response Rate | 8 weeks
  Objective Response Rate as determined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1 and iRECIST
Progression-free survival (PFS) | 5 years
  PFS is measured from the start of treatment to the time of progression or death, whichever occurs first while on the study.
Overall Survival (OS) | 5 years
  OS is defined as the time from Cycle 1 Day1 to death due to any cause.
Duration of Response (DOR) | 5 years
  DOR as determined by RECIST criteria version 1.1 and iRECIST

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - CIP Centro Integrado de Pesquisa / Hospital de Base / Fundação Faculdade de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Instituto do Cancer do Estado de São Paulo (ICESP), São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No